CLINICAL TRIAL: NCT00265746
Title: Program for the Prevention of Diabetes Mellitus Development in Women Who Had Already Experienced A Gestational Diabetes. Evaluation of the Efficacy of the Life-style Modification and the Life-style Modification in Conjunction With Metformin, in the Prevention of Diabetes Mellitus Development in a Population of Women Who Had Expired a Gestational Diabetes - a Multicenter, Randomized, Double Blind Study.
Brief Title: Prevention of Diabetes Mellitus Development in Women Who Had Already Experienced A Gestational Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Medical University Lodz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KBN Nr 2 P05001 28
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: metformin; gestational diabetes; lifestyle
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational | interventions — Metformin; Exercise

INTERVENTIONS:
Drug: Metformin
Behavioral: Lifestyle intervention - diet, physical activity

SUMMARY:
Gestational diabetes is also a strong risk factor for the development of diabetes mellitus at a later stage of life in previous GDM woman. Among all the risk factors of diabetes mellitus, the experience of gestational diabetes is the strongest one. The incidence of various forms of diabetes in this group balances from 10 to 60% over a period from 2 to 10 years.

The aim of this study is a comparison of the efficacy of life style modification and life style modification in conjunction with metformin administration, in a population of women, who had already experienced gestational diabetes.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is one of the most frequent metabolic disorders occurring during pregnancy that complicates both, the course of pregnancy and the delivery and is also responsible for many fetal complications. Gestational diabetes is also a strong risk factor for the development of diabetes mellitus at a later stage of life in previous GDM woman. Among all the risk factors of diabetes mellitus, the experience of gestational diabetes is the strongest one. The incidence of various forms of diabetes in this group balances from 10 to 60% over a period from 2 to 10 years.

Presently, in the literature, there are described new, more efficient methods of diabetes prevention in groups with a high risk of this disorder, which involve both, a modification of the life style and pharmacotherapy. The use of metformin in patients with a impaired glucose tolerance, resulted in a ca. 30% reduction of the diabetes incidence rate.

The aim of this study is a comparison of the efficacy of life style modification and life style modification in conjunction with metformin administration, in a population of women, who had already experienced gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* GDM - experienced during pregnancy (diagnosis of GDM according to WHO-criteria)
* Breast-feeding of the newborn finished (lactation finished)
* Actual BMI >= 25 kg/ m2
* Written consent for participation in the study
* A hitherto prevailing good cooperation with the patient

Exclusion Criteria:

* Cholestasis during the past pregnancy
* Any hepatic diseases in the past (viral hepatitis, toxic hepatic damage,jaundice of unknown etiology)
* Serum ASPAT and/or ALAT level exceeding more than twice normal laboratory values
* Pregnancy planned during the coming two years
* Presence of contradictions for metformin administration according to demands of the Drug Admission Committee in Poland

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11 (Estimated); Primary Completion 2007-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of type 2 diabetes mellitus.

SECONDARY OUTCOMES:
Incidence of IGT

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Cypryk, MD, PhD, Habilitation, Principal Investigator — Medical University in Lodz